CLINICAL TRIAL: NCT06626139
Title: 2 x 2 Factorial, Double-blind, Randomized Trial of 'Set and Setting': a Translational Study in Healthy Volunteers
Brief Title: Investigating the Interaction of Psilocybin and Context of Its Administration in Healthy Volunteers
Acronym: SnS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robin Carhart-Harris, PhD, MA (Other)
Responsible Party: Sponsor-Investigator, Robin Carhart-Harris, PhD, MA, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-38706
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants With Lower-than-average Mental Well-being
Keywords: well-being; psilocybin; psychedelic; neuroimaging; healthy volunteers
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: 2 x 2 Factorial Design Factor 1: Drug (Psilocybin vs Placebo) Factor 2: Context (Context 1 vs Context 2)
Who Masked: Participant, Investigator
Masking Description: Research staff will be masked in reference to the Drug condition but not the Context condition. Participants will be briefed only on the Context condition they are randomized to, and masked in reference to Drug condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Psilocybin C1 (Experimental): Following screening and a baseline assessment visit, healthy volunteers will receive one dose of up to 25mg psilocybin in a context (Context 1) that is hypothesized to modulate acute and post-acute drug effects.
  Interventions: Drug: Psilocybin; Behavioral: Context 1
- Psilocybin C2 (Experimental): Following screening and a baseline assessment visit, healthy volunteers will receive one dose of up to 25mg psilocybin in a context (Context 2) that is hypothesized to modulate acute and post-acute drug effects.
  Interventions: Drug: Psilocybin; Behavioral: Context 2
- Placebo C1 (Placebo Comparator): Following screening and a baseline assessment visit, healthy volunteers will receive one dose of an inactive placebo in a context (Context 1) that is hypothesized to modulate acute and post-acute drug effects.
  Interventions: Behavioral: Context 1; Drug: Placebo
- Placebo C2 (Placebo Comparator): Following screening and a baseline assessment visit, healthy volunteers will receive one dose of an inactive placebo in a context (Context 2) that is hypothesized to modulate acute and post-acute drug effects.
  Interventions: Behavioral: Context 2; Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Healthy participants will receive up to 25 mg psilocybin.
  Arms: Psilocybin C1; Psilocybin C2
Behavioral: Context 1 — Drug administration will take place in a context (Context 1) that is expected to modulate acute and post-acute drug effects.
  Arms: Placebo C1; Psilocybin C1
Behavioral: Context 2 — Drug administration will take place in a context (Context 2) that is expected to modulate acute and post-acute drug effects.
  Arms: Placebo C2; Psilocybin C2
Drug: Placebo — Healthy participants will receive an inactive placebo.
  Arms: Placebo C1; Placebo C2

SUMMARY:
One hundred twenty healthy participants, ages 21 to 70, who experience moderate-to-lower-than-average mental well-being will be evenly randomized into four different study arms, using a 2x2 factorial design. Depending on the study arm, participants will either receive an inactive placebo or up to 25mg psilocybin (oral dose), in one of two set and setting conditions; drug administration contexts that are predicted to modulate drug effects.

The purpose of this study is to evaluate any interaction effects between an oral dose of psilocybin and the surrounding context (set and setting).

DETAILED DESCRIPTION:
Recent research posits that psychedelic medicine is best employed as a combination treatment, i.e., as drug x psychological support or psychotherapy referred to for simplicity as 'psychedelic therapy'. It is assumed that positive outcomes via psychedelic therapy critically depend on a synergistic relationship between drug-induced brain and mind plasticity and supportive contextual factors (Carhart-Harris et al., 2018; Carhart-Harris and Friston, 2019). These contextual factors have been referred to as 'set and setting' (Leary et al., 1963) or 'extrapharmacological'- highlighting elements beyond the drug that contribute to relevant outcomes (Hartogsohn, 2016).

The proposed experiment is a double-blind, randomized between-subjects 2 x 2 factorial study in 120 volunteers who experience low psychological well-being at baseline and have limited prior experience with psychedelics (1:1:1:1, n = 30 per condition). The main aim of the study is to assess the contribution of a select number of pre-defined contextual variables (both 'set' and 'setting') on the nature and trajectory of effects linked to a single dosing session with either psilocybin (oral, 25mg) or placebo (oral, inert).

The study will have four primary outcomes, two pertaining to mental health, namely: changes in psychological well-being - as measured via the Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS), from baseline to 4 weeks post dosing session (primary endpoint) and changes in the Watts Connectedness Scale (WCS) at consistent timepoints. The two primary outcomes indexing the quality of the acute experience will be: Emotional Breakthrough - measured via mean scores on the Emotional Breakthrough Inventory (EBI), and Challenging experience (CE) - defined and measured here as scores on the following four sub-factors of the Challenging Experience Questionnaire (CEQ): fear, insanity, isolation, and paranoia.

ELIGIBILITY:
If you are interested in participating in this study, please follow this link to check your eligibility: https://tiny.ucsf.edu/setsettingscreener

Inclusion Criteria:

Participants will be considered for inclusion if they:

1. Are between 21 and 70 years of age
2. Are fluent in speaking and reading English
3. Are able to swallow pills/capsules
4. If able to become pregnant, must be non-lactating, have a negative pregnancy test at study entry and prior to each Experimental Session and must agree to an adequate form of birth control over the course of the study. Adequate forms of birth control include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Unable to become pregnant is defined as documented hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and/or tubal ligation), permanently sterile by medical device such as Essure, postmenopausal, or assigned male sex at birth.
5. Able and willing to provide informed consent
6. Able and willing to use computers and tablets or phones to enter electronic data
7. Agree to inform the investigators within 48 hours of any new or changed medical conditions.
8. Have an identified support person
9. For those dosed with psilocybin, their prior consent to be accompanied home (or to an otherwise safe destination) by a support person, chosen by them - ahead of time, or by a member of the study team.
10. Willing to provide contact details for a friend or family member, should there be an inability to make direct contact with the participant

Exclusion Criteria:

Participants will be excluded if they:

1. Have a current diagnosed psychiatric disorder that, in the opinion of the study clinician or PI, renders to person psychologically unstable or unduly vulnerable, or interferes with activities of daily living, or could impact attendance at or participation in study activities
2. Have a medically significant condition that renders the person unsuitable for the study
3. Give a positive alcohol breathalyzer test result on any study visit
4. A positive urine drug screen to any excluded substances prior to an Experimental Session, which warrants exclusion based on concerns that it may compromise safety or confound outcomes
5. Are breastfeeding, or have a positive pregnancy test at screening or at any point during the course of the study
6. Systolic and diastolic BP values exceeding 139 SBP and exceeding 89 DBP and heart rate exceeding 90 bpm would result in exclusion from the study.
7. Present with a exceeding 450 msec or with evidence of cardiac damage, ischemia, or heart disease.
8. Have received an investigational drug within 30 days of the screening visit
9. Have an allergy or intolerance to any of the materials contained in either drug product or setting components, such as certain scents.
10. Have MRI contraindications (e.g., metal implants, pacemakers, claustrophobia etc.)
11. Have any current problem which, in the opinion of the investigator or clinician, might interfere with participation.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Challenging Experience Questionnaire (CEQ) subscales score | Eight hours post-dose.
  The Challenging Experience Questionnaire is designed to measure challenging psychological experiences associated with the acute effects of psilocybin. For this study, the combined score across four our of its seven subscales will be used as a primary outcome: Fear, Insanity, Isolation, and Paranoia, excluding Grief, Physical Distress, and Death subscales. Scaled scores range from 0 to 100. Higher scores indicate higher levels of challenging experience (worse outcome).
Change in Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) score from Baseline to 28 days post-dose | Baseline to 28 days post-dose.
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) was developed to enable the monitoring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing. Scores range form 14 to 70. Higher scores indicate higher levels of mental well-being (better outcome).
Change in Watts Connectedness Scale (WCS) scores from Baseline to 28 days post-dose | Baseline to 28 days post-dose.
  The WCS is a 3-dimensional index of felt connectedness that may sensitively measure therapeutically relevant psychological changes post-psychedelic use. Scores range from 0 to 100. Higher scores indicate higher levels of connectedness (better outcome).
Emotional Breakthrough Inventory (EBI) score | Eight hours post-dose.
  The Emotional Breakthrough Inventory was developed to assess emotional breakthrough, an important and distinct component of the acute psychedelic experience. Scores range from 0 to 100. Higher scores indicate higher levels of emotional breakthrough (better outcome).

SECONDARY OUTCOMES:
Changes in resting state BOLD activity viafunctional magnetic resonance imaging (fMRI) | Baseline to 28 days post-dose.
  Assessment parameters include: Eyes-closed resting state fMRI
Changes in BOLD activity during emotional processing via functional magnetic resonance imaging (fMRI) | Baseline to 28 days post-dose.
  Assessment parameters include: BOLD response during an emotional processing task
Changes in white matter organization via magnetic resonance imaging (MRI) | Baseline to 28 days post-dose.
  Assessment parameters include: Diffusion Tensor Imaging (DTI)
Structural brain changes via magnetic resonance imaging (MRI) | Baseline to 28 days post-dose.
  Assessment parameters include: T1- and T2-weighted imaging
Acute Lempel Ziv Complexity (LZC) via Electroencephalography (EEG) | Pre-dose; 2, 4, and 6 hours post-dose
  Electroencephalography is a method to record an electrogram of the spontaneous electrical activity of the brain. Assessment parameters include: Lempel Ziv Complexity (LZC)
Spectral power in traditional frequency bands via Electroencephalography (EEG) | Pre-dose; 2, 4, and 6 hours post-dose
  Electroencephalography is a method to record an electrogram of the spontaneous electrical activity of the brain. Assessment parameters include: Spectral power in traditional frequency bands
Transfer entropy and integrated information via Electroencephalography (EEG) | Pre-dose; 2, 4, and 6 hours post-dose
  Electroencephalography is a method to record an electrogram of the spontaneous electrical activity of the brain. Assessment parameters include: Transfer entropy and integrated information
Synergistic and redundant activity patterns via Electroencephalography (EEG) | Pre-dose; 2, 4, and 6 hours post-dose
  Electroencephalography is a method to record an electrogram of the spontaneous electrical activity of the brain. Analytic approaches include: Partial information decomposition
Travelling waves via Electroencephalography (EEG) | Pre-dose; 2, 4, and 6 hours post-dose
  Electroencephalography is a method to record an electrogram of the spontaneous electrical activity of the brain. Assessment parameters include:
  Travelling waves

CONTACTS AND LOCATIONS:
Overall Officials: Robin Carhart-Harris, PhD, Principal Investigator — University of California, San Francisco; Jennifer Mitchell, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No